CLINICAL TRIAL: NCT06850467
Title: The Impact of Sexual Intercourse on Spontaneous Onset of Labor
Brief Title: Sexual Intercourse on Spontaneous Onset of Labor
Acronym: AchourPrtcol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Medicine of Tunis (Other)
Responsible Party: Principal Investigator, Achour Radhouane, Prof, Faculty of Medicine of Tunis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T00002515
Record Dates: First submitted 2025-02-05; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Sexual Intercourse; Spontaneous Labor
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sexual intercourse protocol (Experimental): Our sample was divided into 2 groups by randomization. The first group (interventional) followed the protocol for 2 weeks. These women were asked to keep a daily diary to record coitus and orgasm activities: the rhythm of sexual intercourse, the nature of the intercourse which must be complete and without a condom.
  Interventions: Behavioral: Sexual intercourse protocol
- Control group (No Intervention): In the control group, sexual intercourse was neither encouraged nor discouraged.

INTERVENTIONS:
Behavioral: Sexual intercourse protocol — The study involved pregnant women who were randomly assigned to 2 groups. The protocol involved engaging in sexual intercourse and nipple stimulation 3 times per day for two consecutive weeks with the consecutive days of sexual intercourse and days of nipple stimulation being different. Patients documented their coital activities as well as the frequency of orgasms in their daily journal. There were no prohibitions regarding or promotions of sexual activities for the control group. The main outcome was the onset of labor, which was defined as the presence of effective uterine contraction with changes of the cervix (Bishop score > 5) without using the induction treatments during protocol time or until 41 weeks of pregnancy.
  Arms: Sexual intercourse protocol

SUMMARY:
Women included in our study were recruited for a randomized trial on the effect of sexual intercourse to promote the onset of spontaneous labor. For this analysis, our sample was divided into two groups by randomization. The first group (experimental) followed the protocol (sexual intercourse 1 day out of 2 alternating with nipple stimulation alone for 15 minutes three times a day) for 2 weeks. In the control group, sexual relations were neither encouraged nor discouraged. Spontaneous labor prior to the date of scheduled labor induction was the primary outcome. We consider that the result is statistically significant differences when P < 0.05.

DETAILED DESCRIPTION:
Participants comprised pregnant women who were receiving prenatal care at the Maternity and Neonatology Center in Tunis (CMNT). This study was a quasi-experimental, comparative, longitudinal, prospective, and monocentric over one year, from September 24, 2021, to September 24, 2022.

Women in the study had to be aged between 18 and 45 years and had to be with uncomplicated singleton pregnancies with gestational age of 37 weeks and above, at low risk for complication, with intact membranes, and in cephalic presentation. Exclusion criteria were pregestational or gestational hypertension, preeclampsia, gestational diabetes, epilepsy in the mother, type 1 or 2 diabetes, contraindications to vaginal delivery, any type of hospitalization, increased surveillance due to suspicion of preterm labor, unexplained vaginal bleeding, sexually transmitted disease, or fetal anomalies.

The study involved pregnant women who were randomly assigned to two groups. The protocol involved engaging in sexual intercourse and nipple stimulation 3 times per day for two consecutive weeks with the consecutive days of sexual intercourse and days of nipple stimulation being different. Patients documented their coital activities as well as the frequency of orgasms in their daily journal. There were no prohibitions regarding or promotions of sexual activities for the control group. The main outcome was the onset of labor, which was defined as the presence of effective uterine contraction with changes of the cervix (Bishop score > 5) without using the induction treatments during protocol time or until 41 weeks of pregnancy.

The subjects were divided into experimental and control groups using simple random sampling. To eliminate group-bias during the allocation, a computer assigned a sequence of random numbers to all the participants. To eliminate selection bias, allocation concealment was ensured by using sequentially numbered, sealed, opaque envelopes which were prepared by an otherwise unrelated third party. Age and parity were considered for stratification of cases and controls to have relatively equal distribution across the groups.

Quantitative data were obtained from the women through self-administered questionnaires which focused on sexual activity during pregnancy and at term. A chi-square test was carried out to determine if there is a significant relationship between sexual intercourse and the incidence of spontaneous onset of labor. Data analysis was performed using SPSS 21 stats software, with a level of significance set at 0.05.

Both the study aim, and protocol were approved by the ethics committee of the Maternity and Neonatology center of Tunis. Informed consent was obtained from all participants. Participants' anonymity and data confidentiality were upheld throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* We included pregnant women (primiparous or multiparous) who presented to the perinatal consultation of the maternity and neonatology center of Tunis. Their pregnancies are evolving singleton, low risk, with intact membranes and cephalic presentation.

Exclusion Criteria:

* The non-inclusion criteria were high-risk pregnancies:

  * pregnancy pathologies: pregnancy-induced hypertension, pre-eclampsia, gestational diabetes, pregnancy-induced cholestasis, IUGR.
  * maternal pathologies: epilepsy, type 1 or 2 diabetes.
  * contraindications to vaginal delivery: placenta previa or accreta, history of two (or more) cesarean sections, breech or transverse presentation.
  * hospitalizations and/or increased monitoring during pregnancy related to a threat of premature delivery, undetermined bleeding, sexually transmitted diseases, fetal pathologies and/or malformations.

Patients who did not follow the protocol for any reason.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 224 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2022-09-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
spontaneous onset of labor | the spontaneous onset of laborduring the protocol (during the 15 days of the protocol) or after the end of the protocol and up to 41 weeks.
  The judgment criterion is the spontaneous onset of labor defined by effective uterine contractions leading to cervical modification (a favorable Bishop score, i.e. greater than 5), and without resorting to treatment (prepedil gel, maturation by probe, cytotec, etc.) during the protocol (during the 15 days of the protocol) or after the end of the protocol and up to 41 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Manouba 2010 Tunisia, Tunis6-TUNISIA, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goodlin RC, Keller DW, Raffin M. Orgasm during late pregnancy. Possible deleterious effects. Obstet Gynecol. 1971 Dec;38(6):916-20. No abstract available. PMID 5125443
- [Background] Tomlinson AJ, Colliver D, Nelson J, Jackson F. Does sexual intercourse at term influence the onset of labour? A survey of attitudes of patients and their partners. J Obstet Gynaecol. 1999 Sep;19(5):466-8. doi: 10.1080/01443619964210. PMID 15512366
- [Background] Singh N, Tripathi R, Mala YM, Yedla N. Breast stimulation in low-risk primigravidas at term: does it aid in spontaneous onset of labour and vaginal delivery? A pilot study. Biomed Res Int. 2014;2014:695037. doi: 10.1155/2014/695037. Epub 2014 Nov 27. PMID 25525601
- [Background] Di Lieto A, Miranda L, Ardito P, Favale P, Albano G. Changes in the Bishop score induced by manual nipple stimulation. A cross-over randomized study. Clin Exp Obstet Gynecol. 1989;16(1):26-9. PMID 2713990
- [Background] Adewole IF, Franklin O, Matiluko AA. Cervical ripening and induction of labour by breast stimulation. Afr J Med Med Sci. 1993 Dec;22(4):81-5. PMID 7839936
- [Background] Salmon YM, Kee WH, Tan SL, Jen SW. Cervical ripening by breast stimulation. Obstet Gynecol. 1986 Jan;67(1):21-4. PMID 3940333
- [Background] Kurt B, Demirel G, Caglayan IS, Doganer A. The Effect on the Birth Process of Endogenous Oxytocin Release Via Coitus at Home in Pregnant Women in the Latent Phase. Z Geburtshilfe Neonatol. 2023 Apr;227(2):134-140. doi: 10.1055/a-2019-5031. Epub 2023 Feb 20. PMID 36808611
- [Background] Foumane P, Mboudou ET, Sama JD, Baba S, Enama Mbatsogo BA, Ngwana L. Sexual activity during pregnancy and prognosis of labor in Cameroonian women: a cohort study. J Matern Fetal Neonatal Med. 2014 Sep;27(13):1305-8. doi: 10.3109/14767058.2013.856412. Epub 2013 Nov 13. PMID 24134484
- [Background] Castro C, Afonso M, Carvalho R, Clode N, Graca LM. Effect of vaginal intercourse on spontaneous labor at term: a randomized controlled trial. Arch Gynecol Obstet. 2014 Dec;290(6):1121-5. doi: 10.1007/s00404-014-3343-0. Epub 2014 Jul 18. PMID 25033717
- [Background] Carbone L, De Vivo V, Saccone G, D'Antonio F, Mercorio A, Raffone A, Arduino B, D'Alessandro P, Sarno L, Conforti A, Maruotti GM, Alviggi C, Zullo F. Sexual Intercourse for Induction of Spontaneous Onset of Labor: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Sex Med. 2019 Nov;16(11):1787-1795. doi: 10.1016/j.jsxm.2019.08.002. Epub 2019 Sep 11. PMID 31521572
- [Background] Tan PC, Yow CM, Omar SZ. Effect of coital activity on onset of labor in women scheduled for labor induction: a randomized controlled trial. Obstet Gynecol. 2007 Oct;110(4):820-6. doi: 10.1097/01.AOG.0000267201.70965.ec. PMID 17906015
- [Background] Tan PC, Yow CM, Omar SZ. Coitus and orgasm at term: effect on spontaneous labour and pregnancy outcome. Singapore Med J. 2009 Nov;50(11):1062-7. PMID 19960160
- [Background] Grivell RM, Reilly AJ, Oakey H, Chan A, Dodd JM. Maternal and neonatal outcomes following induction of labor: a cohort study. Acta Obstet Gynecol Scand. 2012 Feb;91(2):198-203. doi: 10.1111/j.1600-0412.2011.01298.x. Epub 2011 Nov 15. PMID 21995778
- [Background] Kiesewetter B, Lehner R. Maternal outcome monitoring: induction of labor versus spontaneous onset of labor-a retrospective data analysis. Arch Gynecol Obstet. 2012 Jul;286(1):37-41. doi: 10.1007/s00404-012-2239-0. PMID 22298204
- [Background] Christensson K, Nilsson BA, Stock S, Matthiesen AS, Uvnas-Moberg K. Effect of nipple stimulation on uterine activity and on plasma levels of oxytocin in full term, healthy, pregnant women. Acta Obstet Gynecol Scand. 1989;68(3):205-10. doi: 10.3109/00016348909020990. PMID 2618602
- [Background] Kafaei Atrian M, Sadat Z, Rasolzadeh Bidgoly M, Abbaszadeh F, Asghari Jafarabadi M. The association of sexual intercourse during pregnancy with labor onset. Iran Red Crescent Med J. 2014 Dec 26;17(1):e16465. doi: 10.5812/ircmj.16465. eCollection 2015 Jan. PMID 25763253
- [Background] Templeton AA, Cooper I, Kelly RW. Prostaglandin concentrations in the semen of fertile men. J Reprod Fertil. 1978 Jan;52(1):147-50. doi: 10.1530/jrf.0.0520147. PMID 621688